## ÇALIŞMA PROTOKOLÜ

**Çalışmanın adı:** Obez hastalarda zor entübasyonu ve zor maske ventilasyonunu tahmin edebilmede boyun çevresinin çene-ense çevresine oranının diğer ölçümlerle karşılaştırılması.

Çalışmanın Önemi ve Amacı: Zor hava yolunun uygun şekilde yönetimi, anestezi ile ilişkili mortalite ve morbiditenin önlenmesinde önemli bir yer teşkil eder. Zor laringoskopinin prevalansının % 1.5 ile % 20 arasında değiştiği bildirilmiştir ve varlığını tahmin etmek için çeşitli fizik muayene testleri kullanılmaktadır[1]. Havayolunun değerlendirilmesinde mallampati skorlaması,tiromental mesafe, ağız açıklığı, sternomental mesafe, boyun çevresi ölçümü ve üst dudak ısırma testi gibi çeşitli yöntemler kullanılmaktadır [2]. Multifaktöriyel indeksler tekil ölçümlerden biraz daha iyi performans gösterirken, tek başına hiçbir anatomik ölçümün, zor laringoskopinin ve zor entübasyonun öngörülmesi için yüksek bir doğruluğa sahip olduğu bildirilmemiştir. Zor hava yolunun öngörülmesinde birçok yeni yöntemin kullanılması önerilmiştir. Tiromental yükseklik ölçümü, boyun çevresinin ölçümü ve boyun çevresinin tiromental mesafeye oranının ölçümü yeni önerilen yöntemlerdendir ve zor hava yollarının tahmininde başarılı olduğu bildirilmektedir [3].

Çok sayıda obez hasta günlük olarak elektif ve acil operasyonlar geçirmektedir. Hem zor maske ventilasyonu hem de zor entübasyon ile karakterize zor hava yolları, obez hastalarda sıkça görülmektedir. Zor havayolunun önceden tahmin edilebilmesi ve gerekli olan ileri teknolojik ekipmanların önceden hazırlanması, zor havayolunun yönetimini kolaylaştıabilir ve zor havayolu ile ilişkili mortalite ve morbiditeyi azaltabilir. Birçok çalışma, obezite veya morbid obezite ile zor entübasyon arasında bir ilişki olduğunu göstermiştir[4]. Bir meta-analiz, morbid obez hastalarda normal kilolu hastalardan 3 kat daha zor entübasyon olasılığını bildirmiştir [5]. Mallampati skorunun veya artan boyun çevresinin (BÇ) özellikle obez hastalarda zor entübasyonla ilişkili olduğu bildirilmektedir [4,6].

Tiromental yükseklik ve boyun çevresinin ölçümünün erişkin hasta populasyonunda zor havayollarının tahmininde başarılı olduğu gösterilmiştir[3,7]. Ancak obez hastalarda artmış çene altı yağ dokusu nedeniyle bu yöntemlerin yanıltıcı olabileceğini ve boyun çevresinin çene-ense çevresine oranının zor entübasyonu ve zor maske ventilasyonunu ön görmede daha başarılı olabileceğini düşünmekteyiz ve bu konuda çalışma bulunmamaktadır. Amacımız obez hastaların zor havayolu değerlendirmesinde; tiromental yükseklik ölçümünün, boyun çevresinin ölçümünün ve çene-ense çevresinin boyun çevresine oranının zor maske ventilasyonu ve zor entübasyonu öngörüsünü değerlendirmektir.

Gereç ve Yöntem: Trakeal entübasyon gerektiren elektif cerrahi geçirecek, 18 yaş üstü, Vücut Kitle İndeksi (VKİ) en az 30 olan obez hastalar değerlendirmeye alınacak. Servikal omurga anomalisi, acil durum prosedürleri, bilinen zor entübasyon ve planlı uyanık entübasyon olan ve sakallı olan hastalar çalışma dışı bırakılacak. Hastalar ameliyat öncesi preop alanda anestezi uzmanı tarafından değerlendirilecek. Yaş, Cinsiyet, Amerikan Anestezistler Derneği (ASA) fiziksel durumu, horlama öyküsü, obstrüktif uyku apne Sendromu (OSAS) ve sürekli pozitif hava yolu basıncı (CPAP) cihazı kullanımı dahil olmak üzere tam bir tıbbi anamnez alınacak. Hastaların fizik muayenesinde boy, kilo ve sakal varlığı kaydedilecek. VKİ, boy ve kilo ölçümleri kullanılarak hesaplanacak. Mallampati skoru, üst dudak ısırma, kesici dişler arası mesafe, tiromental mesafe, sternomental mesafe ve tiromental yükseklik dahil olmak üzere hava yolu ölçüm parametreleri kaydedilecek. Bir mezura kullanılarak, nötr pozisyonda tiroid kıkırdak seviyesinden boyun çevresi ve mentum seviyesinden çene-ense çevresi ölçülecek. Boyun

çevresinin tiromental mesafeye oranı ve boyun çevresinin çene-ense çevresine oranı bu ölçümlerden hesaplanacak. Ameliyat öncesi incelemeler kurumun standart uygulamasına göre yapılacak ve ek tetkik istenmeyecek. Eğitimli bir araştırma görevlisi tüm preoperatif hasta verilerini kaydedecek. İndüksiyon öncesi hastalara, trakeal entübasyonu kolaylaştırmak için ameliyat masasında rampa pozisyonu verilecek. Hastalara elektrokardiyogram, pulse oksimetri ve non-invaziv arteriyel kan basıncı monitörizasyonu vapılacak. En az 3 dakika süreyle preoksijenasyon yapılacak. Anestezi indüksiyonu ve idamesi kurumumuzun standart protokolü uygulanarak gerçekleştirilecek. Her vakada aynı anestezist yer alacak ve havayolu yönetiminde en az 2 yıllık klinik deneyime sahip olacak. Maske ventilasyonu, katılan anestezi uzmanının belirlediği şekilde uygun boyutta bir yüz maskesi kullanılarak yapılacak. Maske havalandırması, Han tarafından açıklanan yönteme göre derecelendirilecek. Normal etkili maske ventilasyonu Grade 1, oral airway veya baska bir yardımcı alet ihtiyacı varsa Grade 2, Akciğerlerin ventilasyonunun oksijenlenmeyi sürdürmek için yetersiz olduğu veya maske ventilasyonunun dengesiz olduğu veya ventilasyon için iki kişiye ihtiyaç duyulduğu derece zor Grade 3, Son olarak imkansız ventilasyon Grade 4 olarak derecelendirilecek. Bu çalışmada zor maske ventilasyonu, maske ventilasyonu Grade 3 veya Grade 4 olarak tanımlanacak. Yeterli kas gevşemesi sağlandıktan sonra, uygun boyutta bir Macintosh bleydi ile doğrudan laringoskopi kullanılarak trakeal entübasyon gerçekleştirilecek. Entübasyon sırasında zorluklarla karşılaşılırsa, yardımcı aletlerin veya alternatiflerin kullanımına izin verilecek. Yedi değişkene dayalı Zor Entübasyon Ölçeği (Intubation Difficulty Scale:IDS) kullanılacak: entübasyon girişimi sayısı, ek operatörler, alternatif entübasyon teknikleri, vokal kord pozisyonu, Cormack ve Lehane'nin laringoskopik görünüm için sınıflandırılması, dış laringeal basınca ihtiyaç ve laringoskopla kaldırma kuvveti. Yedi değişkenin tümü değerlendirilecek ve IDS hesaplananacak. Bu çalışmada, IDS 5'in altındaki herhangi bir değer kolay kabul edilecek. Trakeal entübasyon, uygun bir kapnograf dalga formu ile kanıtlandığında ve oskültasyonla her iki akciğer sesleri eşit duyulduğunda başarıyla tamamlandı kabul edilecek.

**Bakılacak parametreler:** Yaş, Boy, Kilo, VKİ, sakal varlığı, Mallampati skoru, Ağız açıklığı, kesici dişler arası mesafe, Tiromental mesafe, Sternomental mesafe, Tiromental yükseklik, üst dudak ısırma, Boyun çevresi, Çene-ense çevresi,Boyun çevresinin tiromental mesafeye oranı, boyun çevresinin çene-ense çevresine oranı, Maske ventilasyon derecelendirmesi, Cormack ve lehane skoru, Zor entübasyon ölçeği **Çalışmaya dahil olma kriteri**: 18 yaş üstü Trakeal entübasyon gerektiren elektif cerrahi geçirecek BMI'si en az 30 olan obez hastalar

Çalışmaya Alınmama Kriterleri: Servikal omurga anomalisi, acil durum prosedürleri, bilinen zor entübasyon ve planlı uyanık entübasyon olan hastalar, sakallı hastalar

Öngörülen Çalışma Süresi: 6 ay

Çalışmanın Orjinalliği: : boyun çevresinin çene-ense çevresine oranının obez hastalarda zor

entübasyonu tahmin etme gücü hakkında çalışma olmaması.

**İstatistiksel Yöntem**: Güç analizi PASS11 (hintze J. NCSS, LLC. Keysville, Utah, USA) programı ile yapıldı. Daha önce boyun çevresinin çene-ense çevresine oranına bakılan literatürde çalışma bulunmadığından dolayı çalışmanın güç analizi yapılırken Kim ve ark. yaptıkları çalışmadaki boyun çevresinin sternomental uzaklığa olan oranı referans olarak alınmıştır (8). Buna göre %90 güç ve 0.05 alfa hata düzeyinde anlamlı

farklılık elde etmek adına en az 12 kolay entübasyon (IDS<5), en az 12 de zor entübasyon hastası (IDS≥5) çalışmaya dahil edilecektir (Ek-1). Obez hastalarda zor entübasyon oranı kolay entübasyon oranına göre daha düşük olduğu için en az 12 zor entübasyon hastası olana kadar tüm obez hastalar çalışmaya alınacak.

Frekans dağılımları sayı ve yüzde, sürekli değişkenler ortalama±standart sapma ve/veya median (minimum-maksimum) şeklinde ifade edilecektir. Sürekli değişkenlerin normal dağılıma uygunlukları Kolmogorov Simirnov Uyum İyiliği Testi ile analiz edilecek, normal dağılıma uyuyor ise T-Testi, uymuyorsa Mann Whitney U Testi kullanılacaktır. Tekrarlayan verilerin analizi Friedman Testi ve Wilcoxon Sıralı İşaret Testi ile yapılacaktır. Kesikli değişkenler arasındaki ilişki Ki-kare Testi ile değerlendirilecektir. Verilerin analizinde İBM SPSS versiyon 24.0 İstatistik Programı kullanılacak, istatistiksel anlamlılık düzeyi p<0,05 olarak ele alınacaktır.

## Kaynaklar:

- 1- Rose DK, Cohen MM. The airway: problems and predictions in 18,500 patients. Can J Anaesth 1994;41:372–83
- 2- Khan ZH,Mohammadi M, RasouliMR, Farrokhnia F, Khan RH. The diagnostic value of the upper lip bite test combined with sternomental distance, thyromental distance, and interincisor distance for prediction of easy laryngoscopy and intubation: a prospective study. Anesth Analg 2009;109:822-4.
- 3- Etezadi F, Ahangari A, Shokri H, Najafi A, Khajavi MR, Daghigh M, et al. Thyromental height: a new clinical test for prediction of difficult laryngoscopy. Anesth Analg 2013;117:1347-51.
- 4- Juvin P, Lavaut E, Dupont H, et al. Difficult tracheal intubation is more common in obese than in lean patients. Anesth Analg 2003; 97:595–600.
- 5- Shiga T, Wajima Z, Inoue T, Sakamoto A. Predicting difficult intubation in apparently normal patients: a meta-analysis of bedside screening test performance. Anesthesiology 2005; 103:429–437.
- 6- Brodsky J, Lemmens H, Brock-Utne J, Vierra M, Saidman L. Morbid obesity and tracheal intubation. Anesth Analg 2002; 94: 732–6
- 7- Neck circumference as a predictor of difficult intubation and difficult mask ventilation in morbidly obese patients A prospective observational study. Waleed Riad, Mercedeh N. Vaez, Ravi Raveendran, Amanda D. Tam, Fayez A. Quereshy, Frances Chung and David T. Wong Eur J Anaesthesiol 2016; 33:244–249
- 8- Kim WH, Ahn HJ, Lee CJ, Shin BS, Ko JS, Choi SJ, Ryu SA. Neck circumference to thyromental distance ratio: a new predictor of difficult intubation in obese patients. *Br J Anaesth*. 2011;106(5):743-748. doi:10.1093/bja/aer024